CLINICAL TRIAL: NCT00794456
Title: Double Blind, Randomized Study, Controlled by Valeriana Officinalis, of Association of Passiflora Incarnata L; Crataegus Oxyacantha L and Salix Alba L. on Patients With Mild and Moderate Anxiety
Brief Title: Association of Passiflora Incarnata L; Crataegus Oxyacantha L and Salix Alba L. on Mild and Moderate Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marjan Industria e Comercio ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MJ 3002-08
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Anxiety Disorder
Keywords: Passiflora; Crataegus; Herbal; Valeriana; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — crataegus extract; willow bark extract; Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Association of Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L.
  Interventions: Drug: Passiflora ; Crataegus and Salix
- 2 (Active Comparator): Valeriana officinalis 50 mg
  Interventions: Drug: Valeriana

INTERVENTIONS:
Drug: Passiflora ; Crataegus and Salix — 1 tablet PO twice a day
  Other Names: Pasalix
  Arms: 1
Drug: Valeriana — 1 tablet PO twice a day
  Other Names: Valeriana officinalis 50 mg
  Arms: 2

SUMMARY:
Phase III, multicentric, double blind, randomized study, controlled by Valeriana officinalis for evaluating the efficacy of association of Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L. on mild and moderate anxiety. The treatment period will last 6 weeks and be followed by a post treatment visit.

Hamilton anxiety scale will be used to assess anxiety.

DETAILED DESCRIPTION:
Passiflora incarnata L; Crataegus Oxyacantha L are plant-derived treatment widely used to treat anxiety disorders. This study will compare the association of Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L for the treatment of mild and moderate anxiety. 150 participants will be randomly assigned to receive the association of Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L. or Valeriana officinalis for 6 weeks. A post treatment visit will be done 2 weeks for safety evaluation.

Primary outcome: Hamilton anxiety (HAM-A) scale Secondary outcome: Insomnia quality index, Global clinical impression and patients global evaluation scales.

Side effects will be monitorized throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* generalized anxiety disorder
* HAM-A scale < 17 and > 30

Exclusion Criteria:

* hypersensibility to any component
* patients with depression, schizophrenia ou suicidal ideas
* pregnant ou lactating
* heart, liver, lung or kidney important condition
* use of digitalis, AAS, anticoagulants agents, drugs with sedative or antidepressant action
* psychotherapy
* drug or alcohol dependence
* gastrointestinal ulcer history
* hyperthyroidism
* neoplasia
* coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hamilton anxiety scale | 6 weeks

SECONDARY OUTCOMES:
Insomnia gravity index; global clinical impression; patients global evaluation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabete A Moraes, MD, Principal Investigator — Federal University of Ceará; Antonio C Lopes, Phd, Principal Investigator — Federal University of Sao Paulo - UNIFESP / DPDM - Associação Paulista para o Desenvolvimento da Medicina - Hospital São Paulo
Locations (2):
- Brazil (2):
  - Unidade de Farmacologia Clínica - UNIFAC, Fortaleza, Ceará
  - SPDM - Associação Paulista para o Desenvolvimento da Medicina - Hospital São Paulo, São Paulo, São Paulo